CLINICAL TRIAL: NCT06250062
Title: A Phase II, Randomized, Double-blind, Placebo-controlled , Multicenter Study to Evaluate the Preliminary Efficacy and Safety of Subcutaneous Injection of Recombinant Humanized Anti-IL-17A Monoclonal Antibody（JS005） in Adult Patients With Active Ankylosing Spondylitis
Brief Title: A Clinical Study of JS005 in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS005-006-Ⅱ-AS
Record Dates: First submitted 2024-01-09; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo（JS005） (Experimental)
  Interventions: Drug: Placebo（JS005）
- Recombinant humanized IL-17A Monoclonal Antibody（JS005）150mg (Experimental)
  Interventions: Drug: Recombinant humanized IL-17A Monoclonal Antibody（JS005）; Drug: Placebo（JS005）
- Recombinant humanized IL-17A Monoclonal Antibody（JS005）300mg (Experimental)
  Interventions: Drug: Recombinant humanized IL-17A Monoclonal Antibody（JS005）; Drug: Placebo（JS005）

INTERVENTIONS:
Drug: Recombinant humanized IL-17A Monoclonal Antibody（JS005） — Injection
  Arms: Recombinant humanized IL-17A Monoclonal Antibody（JS005）150mg; Recombinant humanized IL-17A Monoclonal Antibody（JS005）300mg
Drug: Placebo（JS005） — Injection

SUMMARY:
This is a multicentre, randomized, double-blind, parallel, placebo-controlled Phase II clinical study of 261 adults with active ankylosing spondylitis to evaluate the efficacy and safety of JS005 in the treatment of active ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily particpate in this clinical study and sign the informed consent form.
2. Male and female patients aged 18-75 years at the time of screening (both inclusive)
3. Meet the diagnosis of active Ankylosing Spondylitis(AS), have a record of radiological evidence consistent with the Modified New York Classification Criteria for ankylosing spondylitis as revised in 1984 4. Diagnosis of active AS (active AS is defined as: BASDAI >= 4, total back pain score >=4, and BASDAI second question spinal pain score >=4)

Exclusion Criteria:

1. Pregnant or lactating women.
2. Active diseases that may confound the evaluation of JS005: other autoimmune inflammatory diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, sarcoidosis, vasculitis, etc.) or chronic pain other than ankylosing spondylitis (including but not limited to fibromyalgia, osteoarthritis, etc.).

4. Active inflammatory bowel disease within 6 months prior to randomization. 5. Recurrent anterior uveitis or acute anterior uveitis within the last 4 weeks prior to randomization.

6. History or evidence of active or latent tuberculosis (TB), defined as a positive interferon gamma release assay (IGRA) or purified protein derivative (PPD) at the time of screening. 7. Positive hepatitis B virus test result 8. Prior exposure to JS005 or any other biologic that directly targets IL-17 or the IL-17 receptor.

9. use of >= 2 TNF-α inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-02-26 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of SpondyloArthritis International Society criteria (ASAS）40 | 16 weeks
  Proportion of subjects meeting Assessment of SpondyloArthritis International Society criteria (ASAS）40 response criteria at week 16.

SECONDARY OUTCOMES:
Assessment of SpondyloArthritis International Society criteria (ASAS）40 | 32 weeks
  Proportion of subjects meeting Assessment of SpondyloArthritis International Society criteria (ASAS）40 response criteria at week 32.
Assessment of SpondyloArthritis International Society criteria (ASAS）20 | 16 weeks and 32 weeks
  Proportion of subjects meeting Assessment of SpondyloArthritis International Society criteria (ASAS）20 response criteria at weeks 16 and 32.
Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) | 16 weeks and 32 weeks
  Changes in ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) from baseline at weeks 16 and 32
Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) <2.1 | 16 weeks and 32 weeks
  Proportion of subjects with ASDAS-CRP less than 2.1 at weeks 16 and 32.
Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) ≥ 1.1 | 16 weeks and 32 weeks
  The proportion of subjects with Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) change of 1.1 or greater from baselinat weeks 16 and 32.
Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) ≥ 2.0 | 16 weeks and 32 weeks
  The proportion of subjects with Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) change of 2.0 or greater from baselinat weeks 16 and 32.
Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) < 1.3 | 16 weeks and 32 weeks
  Proportion of subjects with Ankylosing spondylitis disease activity score C-Reactive Protein (ASDAS-CRP) less than 1.3 at weeks 16 and 32
Assessment of SpondyloArthritis International Society criteria (ASAS) partial remission | 16 weeks and 32 weeks
  Proportion of subjects who achieved partial remission of Assessment of SpondyloArthritis International Society criteria (ASAS) at weeks 16 and 32
Pharmacokinetic(PK) | 40 weeks
  To evaluate the pharmacokinetic characteristics of JS005: blood concentration of JS005
Immunogenicity | 40 weeks
  The immunogenicity of JS005 was assessed by the positive incidence and titer of drug-resistant antibodies (ADA) and the incidence of neutralizing antibodies (NAb), if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Huji Xu, PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (38):
- China (38):
  - Beijing Chao-yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Jilin Province People's Hospital, Jilin, Changchun
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southren Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Nanyang Central Hospital, Nanyang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - The First Affiliated Hospital of Baotou Medical University, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First People's Hospital of Jiujiang City, Jiujiang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Bethune First Hospital Of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No